CLINICAL TRIAL: NCT06586567
Title: Association of Helicobacter Pylori Infection With Disease Activity in Systemic Lupus Erythrematosis and Rheumatoid Arthritis
Brief Title: H-pylori Infection With Disease Activity in Systemic Lupus Erythematosus and Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Mostafa Mohamed Ahmed, Principal Investigator, Assiut University
Other Study IDs: H pylori and SlE and RA
Record Dates: First submitted 2024-02-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Restraint, Physical; Blood Cell Count; Blood Urea Nitrogen; Gastroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 (SLE group):: 50 patients fulfilling the1997 revised American Collage of Rheumatology classification criteria for SLE according to (Hochberg, 1997)., and h_pylori positive
  Interventions: Other: Full history , clinical examination, assesment of disease activity ,Laboratory investigations ( CBC , ESR, CRP Serum creatinine and blood urea, Random plas
- Group 2 (RA group):: 50 RA patients diagnosed according to the American college of rheumatology (ACR)-EULAR RA classification criteria 2010. And H_pylori positive
  Interventions: Other: Full history , clinical examination, assesment of disease activity ,Laboratory investigations ( CBC , ESR, CRP Serum creatinine and blood urea, Random plas
- Group 3: 50 heqlthy age and sex matched adults were selected as control group
  Interventions: Other: Full history , clinical examination, assesment of disease activity ,Laboratory investigations ( CBC , ESR, CRP Serum creatinine and blood urea, Random plas

INTERVENTIONS:
Other: Full history , clinical examination, assesment of disease activity ,Laboratory investigations ( CBC , ESR, CRP Serum creatinine and blood urea, Random plas — 2. Complete clinical examination 3. Assessment of disease activity
  The following disease activity parameters were used to assess the current activity of each disease:
  * Disease activity score (DAS-28) for patients with RA.
  * SLE disease activity scale (SLEDAI) for patients with SLE. 4. Laboratory investigations: Complete blood count (CBC) Erythrocyte sedimentation rate (ESR). C-reactive protein (CRP) Serum creatinine and blood urea Random plasma glucose level Liver function tests Complete urine analysis. 24 hours urinary protein (g/day) 24 hours creatinine clearance Uric acid Complement 3& 4. Antinuclear antibody (ANA) Anti-dsDNA antibody Estimation of H.Pylori
  Other Names: Upper endoscopy

SUMMARY:
To find the relation of Helicobacter pylori with disease activity in SLE and RA

DETAILED DESCRIPTION:
H. pylori is a widespread, spiral-shaped, flagellated Gram-negative bacterium usually infects the gastric mucosa.Its seropositivity increases with age as it affects about eighty percent of the middle-aged adults in the developing countries and about twenty-five to fifty percent in the western populations.The relation between infection and autoimmune diseases has been previously investigated. Many Gram-negative bacteria as salmonella, shigella, and chlamydia were confirmed to be associated with the development of reactive arthritis.These bacteria have been found to stimulate the host immune response due to the presence of lipopolysaccharides and other antigenic molecules that can cause inflammation.It has been previously hypothesized that H. pylori can induce such immune host response through many mechanisms as the molecular mimicry and antigenic similarity, disruption of the tolerogenic immune response, and activation of the polyclonal lymphocytes leading ultimately to the imbalance between T regulatory/Th17 cells in addition to the induction of autoantibody production

ELIGIBILITY:
Inclusion Criteria:

1. patients with SLE and RA who were admitted to Rheumatology unit in Internal medicine department, Assuit University Hospital will be enrolled in this study

Exclusion Criteria:

* Any patient or control known to have treatment for H. pylori or taking antibiotic treatment for the previous three months 2- Patients receiving biologic therapy 3-Patients known to have diabetes mellitus, autoimmune thyroid disease or autoimmune hepatitis or any other autoimmune

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient of RA and SLE above the age of 18 yrs Presented with hyplori infection
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-04 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of activity of SLE and RA after treatment of H Pylori infection | 2 years
  Prevalence of activity of SLE and RA after treatment of H Pylori infection

REFERENCES:
- [Background] Fontes M. Purification and properties of acid phosphatases isolated from Owenia fusiformis. Biochimie. 1976;58(10):1155-8. doi: 10.1016/s0300-9084(76)80113-7. PMID 12839
- [Background] Hahn P, Vikterlof KJ, Rydman H, Beckman KW, Blom O. The value of whole body bone scan in the pre-operative assessment in carcinoma of the breast. Eur J Nucl Med. 1979 Jun 1;4(3):207-10. doi: 10.1007/BF00620487. PMID 115691
- [Background] Zanchetti A, Stella A, Leonetti G, Morganti A, Terzoli L. Control of renin release: a review of experimental evidence and clinical implications. Am J Cardiol. 1976 Mar 31;37(4):675-91. doi: 10.1016/0002-9149(76)90413-6. PMID 3964